CLINICAL TRIAL: NCT05110638
Title: A Phase 1, Open-Label Study Evaluating the Pharmacokinetics, Absorption, Safety and Tolerability With Maximal Use of SKX-16 (Luliconazole 10% Solution) in Subjects With Moderate to Severe Distal Subungual Onychomycosis
Brief Title: Safety and Tolerability Study of SKX-16 in Subjects With Moderate to Severe Distal Subungual Onychomycosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SATO Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKX16A01
Record Dates: First submitted 2021-07-25; First posted 2021-11-08 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Onychomycosis of Toenail
Keywords: Onychomycosis
MeSH Terms: conditions — Onychomycosis | interventions — luliconazole; Solutions

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SKX-16 (Luliconazole 10% Solution) (Experimental)
  Interventions: Drug: SKX-16 (Luliconazole 10% Solution)

INTERVENTIONS:
Drug: SKX-16 (Luliconazole 10% Solution) — SKX-16 (Luliconazole 10% Solution) will be applied to each toenail and periungual areas once daily for 29 days such that there is sufficient quantity of solution to treat all toenails. All ten toes will be treated regardless of whether affected. The applications will occur in the clinic and be applied by study personnel. The nails will remain exposed until the applied solution dries.

SUMMARY:
This study is being conducted to determine the pharmacokinetics, systemic exposure, safety and tolerability after daily topical application of SKX-16 (Luliconazole 10% Solution) for duration of 29 days in a maximal use setting in adults with moderate to severe distal subungual onychomycosis of the toenails.

DETAILED DESCRIPTION:
Subjects in this open-label study will receive once daily, topical applications of SKX-16 (Luliconazole 10% Solution) in the clinic for 29 days. Subjects will be followed for seven days after the last application (Day 29).

Subjects will be admitted into the study after written informed consent has been obtained and all inclusion/exclusion criteria have been met.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects demonstrate ability and willingness to sign a written informed consent.
2. Subjects of either gender, any race and between the ages of 18 and 65 inclusive.
3. Subjects must have ten toes.
4. Subjects with a clinical diagnosis of distal subungual onychomycosis involving both great toenails and ≥ 50% of at least one of the great toenails, as determined by visual inspection after the nail is trimmed.
5. In addition to both great toenails, subjects must have at least four additional toenails with clinical diagnosis of distal subungual onychomycosis.
6. Subjects must have a mycological diagnosis of distal subungual onychomycosis: fungal hyphae on KOH wet mount and positive fungal culture for dermatophyte (microbial infection with fungus belonging to the genus Trichophyton, Microsporum, Epidermophyton) from at least one great toenail.
7. Subjects must have normal renal function as measured by serum creatinine < ULN.
8. Subjects must have normal hepatic function as measured by aspartate aminotransferase (AST/SGOT), alanine aminotransferase (ALT/SGPT), and total bilirubin < ULN.
9. Females of child-bearing potential (FOCBP) must have a negative urine pregnancy test and must agree to use a highly effective form of contraception or abstinence and be willing to remain on that same method of birth control throughout the study.
10. Subjects must be free of any disease that in the Investigator's opinion might interfere with the study evaluations or jeopardize the subject's safety.
11. Subject must be able to communicate, be able to understand the study procedures, and be willing to comply with the study requirements.

Exclusion Criteria:

1. Subjects with a history of intolerance or hypersensitivity to imidazole compounds or the inactive components of the solution.
2. Subjects with an abnormal ECG morphology and/or a QTcF interval > 450 ms for males and >470 ms for females.
3. Subjects with any history of cardiac disease or cardiac rhythm abnormalities.
4. Subjects with symptomatic tinea pedis at baseline.
5. Subjects unwilling to refrain from the use of nail cosmetics including nail lacquers from the Screening visit until the end of the study.
6. Female subjects who are pregnant and/or nursing or planning a pregnancy during the course of the trial.
7. Concomitant use of any drugs that are CYP3A and CYP2C19 substrates with QT interval prolongation potential.
8. Subjects who have not undergone the specified washout period(s) prior to Baseline visit (Day 1) for the following topical preparations, or subjects requiring the concurrent use of any of the following topical medications: Topical antifungal applied to the feet, drugs that contain luliconazole, anti-inflammatories, corticosteroids or topical immunomodulators.
9. Systemic antifungals for treatment of onychomycosis or any systemic antifungal with known activity against dermatophytes within the previous 12 weeks or 5 half-lives of the drug, whichever is longer.
10. Subjects who have not undergone the specified washout period(s) prior to Baseline (Day 1) for the following systemic medications, or subjects requiring the concurrent use of any of the following systemic medications: Corticosteroids (including intramuscular injections), systemic immunomodulators and drugs that are CYP3A and CYP2C19 substrates
11. Subjects receiving any other treatment/therapy for their onychomycosis not previously mentioned (e.g., laser treatment) who have not undergone a washout period of 4 weeks.
12. Subjects with a history of significant internal disease (including diabetes that is uncontrolled), history or signs of peripheral circulatory insufficiency and/or diabetic neuropathy, recurrent cellulitis or with a life-threatening condition (e.g., autoimmune deficiency syndrome, cancer, unstable angina, or myocardial infarction) as assessed by the Investigator within the last 6 months.
13. Subjects with anatomic abnormalities of the toe(s) and/or toenails, e.g., genetic nail disorders, trauma to the toenail(s).
14. Subjects with a recent history of or currently known to abuse drugs or alcohol.
15. Subjects who have donated or lost a large volume of blood (~500 mL or more), during the 6-week period preceding Baseline visit (Day 1).
16. Subjects who are currently participating in another investigational medication or device study or have participated in a clinical trial within 30 days or 5 half-lives of the test medication (whichever is longer) prior to Baseline visit (Day 1) of this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-12-10 (Estimated); Study Completion 2023-02-22 (Estimated)

PRIMARY OUTCOMES:
PK parameters for the systemic absorption of luliconazole - AUC0-24h | 36 days
  The pharmacokinetics parameter AUC0-24h (the area under the concentration versus time curve measured to the 24 hour time point) will be measured for systemic absorption of luliconazole
PK parameters for the systemic absorption of luliconazole - AUC0-∞ | 36 days
  The pharmacokinetics parameter AUC0-∞ (the area under the concentration versus time curve measured to the end of the sampling period) will be measured for systemic absorption of luliconazole.
PK parameters for the systemic absorption of luliconazole - Cmax | 36 days
  The pharmacokinetics parameter Cmax (the maximum observed concentration over the 0-24 hour interval) will be measured for systemic absorption of luliconazole.
PK parameters for the systemic absorption of luliconazole - Tmax | 36 days
  The pharmacokinetics parameter Tmax (the time to maximum observed concentration over the 0-24 hour interval) will be measured for systemic absorption of luliconazole.
PK parameters for the systemic absorption of luliconazole - t1/2 | 36 days
  The pharmacokinetics parameter t1/2 (the time to maximum observed concentration over the 0-24 hour interval) will be measured for systemic absorption of luliconazole.
PK parameters for the systemic absorption of luliconazole - kel | 36 days
  The pharmacokinetics parameter kel (elimination rate constant) will be measured for systemic absorption of luliconazole.
Safety Assessment - Local Application Site Tolerability Assessment (LASTA) | 36 days
  Evaluation of burning/stinging, pruritus, erythema, and erosion assessed through to Day 29/ET on a scale of 0 to 3 where 0 indicates none and 3 indicates severe.
Safety Assessment - Adverse Events | 36 days
  Subjects will be asked about AEs at each visit; descriptions of AEs will include at minimum: date of onset, date ended, location (whether or not AE is in the treatment area), severity, seriousness, relationship to study drug, and outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Brent Clary, CCRC, Study Chair — Clinical Research Coordinator J&S Studies, Inc.
Locations (1):
- J&S Studies, Inc., College Station, Texas, United States